CLINICAL TRIAL: NCT05344365
Title: An Open-label, Sequential Cohorts, Flexible Dose Study to Evaluate the Tolerability, Safety and Pharmacokinetics of Iloperidone in Elderly Patients With Parkinson's Disease Psychosis (PDP)
Brief Title: A Study to Evaluate Iloperidone for the Treatment of Parkinson's Disease Psychosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated for business reasons; not due to safety or efficacy concerns.
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VP-VYV-683-2301
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease Psychosis
MeSH Terms: interventions — iloperidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iloperidone (Cohort 1) (Experimental)
  Interventions: Drug: Iloperidone
- Iloperidone (Cohort 2) (Experimental)
  Interventions: Drug: Iloperidone

INTERVENTIONS:
Drug: Iloperidone — oral tablet
  Other Names: VYV-683; FANAPT

SUMMARY:
This is an open-label, sequential cohorts, flexible dose study to evaluate the tolerability, safety and pharmacokinetics of iloperidone in elderly patients with Parkinson's disease psychosis (PDP).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide consent and willing to complete all aspects of the study.
* Male or female patients greater or equal to 65 years of age.
* Clinical diagnosis of idiopathic Parkinson's disease with a minimum duration of 1 year
* Psychotic symptoms for at least one month and actively experiencing psychotic symptoms each week during the month prior to screening

Exclusion Criteria:

* History of significant psychotic disorders prior to or concomitantly with the diagnosis of Parkinson's disease including, but not limited to, schizophrenia or bipolar disorder
* Current evidence of a serious and or unstable cardiovascular, respiratory, gastrointestinal, renal, hematologic or other medical disorder, including cancer or malignancies, which would affect the patient's ability to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of iloperidone in patients with Parkinson's disease psychosis. | 8 days and 5 weeks
  As measured by the incidence of adverse events and clinically significant changes in laboratory values, ECG parameters, and vital signs.
Reduction in positive symptoms of Parkinson's disease psychosis. | 8 days and 5 weeks
  As measured by the Scale for the Assessment of Positive Symptoms for Parkinson's Disease Psychosis (SAPS-PD).
Pharmacokinetics of iloperidone and its metabolites following oral treatment with iloperidone. | 8 days and 5 weeks
  As measured by plasma concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, St. Petersburg, Florida, United States